CLINICAL TRIAL: NCT03156010
Title: Oculomotor Assessment of Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Neurolign (Industry); Sync-Think, Inc. (Industry); Oculogica, Inc. (Industry); TBICoE (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. John King, Audiologist, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WRNMMC-2017-0045
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Traumatic Brain Injury
Keywords: oculomotor testing
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: All participants undergo testing with the same three devices. The order of devices will be semi-randomized to eliminate order effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- TBI Group (Other): Subjects with history of TBI will undergo testing with all three devices.
  Interventions: Device: Neuro Kinetics IPAS; Device: Oculogica EyeBox; Device: SyncThink EyeSync Device
- Control Group (Other): Subjects with no history of TBI will undergo testing with all three devices.
  Interventions: Device: Neuro Kinetics IPAS; Device: Oculogica EyeBox; Device: SyncThink EyeSync Device

INTERVENTIONS:
Device: Neuro Kinetics IPAS — Testing with PAS device
Device: Oculogica EyeBox — Testing with Oculogica EyeBox device
Device: SyncThink EyeSync Device — Testing with SyncThink EyeSync device

SUMMARY:
The purpose of the proposed study is to compare the sensitivity and specificity of three oculomotor test devices in normal subjects versus subjects with history of TBI. The study is designed as a prospective research project in which a group of 120 normal controls without a history of TBI will be compared to another group of 120 participants (total of 240) who have a confirmed history of TBI. Each participant will complete the TBI assessment protocol for each of three separate devices (Neuro Kinetics, SyncThink, and Oculogica). The order of the devices will be counter-balanced across participants. Participants will also be screened for vestibular migraine and visual vertigo, which are two conditions that influence oculo-vestibular perception in normal and TBI patients and might influence the results from the three oculomotor devices. Data from each device will be utilized to perform AUC analyses to determine the respective sensitivity and specificity for each.

ELIGIBILITY:
All participants must be DEERS eligible, no exceptions!

Inclusion Criteria:

* Must be between 18 and 45 at time of screening (upper age restriction is to prevent confounding with age-related physiological changes).
* Must be able to provide written informed consent.
* Must be able to read and understand questionnaires and consent forms.
* Must have corrected binocular acuity of at least 20/40 for near distance with or without single-power corrective lenses or contacts and absent of ocular injury or disease.

Control Group - No history of TBI or any history of severe or penetrating TBI

TBI Group - Must have a documented history of a TBI occurring within the last 10 years.

Exclusion Criteria:

* Current or previous neurological disease, including: stroke, congenital brain malformation, degenerative illness such as multiple sclerosis, epilepsy or seizure (other than febrile seizure).
* Current or previous ocular disease/injury, including: Glaucoma or increased pressure in the eyes, structural damage to ocular tract and ocular cortex, etc.
* History of vestibular disorder (e.g., with symptoms of clinical vertigo)
* Binocular vision not correctable to 20/40 for near distance
* Use of tobacco or caffeinated products less than four hours before test session
* Consumption of alcohol within past 24 hours

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) | Single test session (1.5 hours) - all testing performed at time of study enrollment, will be reported at conclusion of data collection as all data is required to generate AUCs.
  Determination of sensitivity/specificity measure for each device using known characteristics of arms (i.e., history of TBI vs no history of TBI)

CONTACTS AND LOCATIONS:
Overall Officials: Louis French, PsyD, Principal Investigator — NICoE
Locations (1):
- National Intrepid Center of Excellence, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. All data from project will be shared in de-identified format as group data, not IPD.